CLINICAL TRIAL: NCT02446106
Title: The Effect of Monosodium L-glutamate (MSG) on Satiety and Energy Intake in Overweight and Obese Women
Brief Title: Monosodium L-glutamate (MSG) on Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajinomoto Co., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 12/NS/0068
Record Dates: First submitted 2015-05-08; First posted 2015-05-18 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Nutrition Intervention
Keywords: Monosodium L-Glutamate (MSG); Satiety; Soups; Energy Intake; Snack Intake
MeSH Terms: interventions — Sodium Glutamate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soup with MSG (Active Comparator): 0.5% MSG incorporated into a soup preload
  Interventions: Dietary Supplement: Soup with MSG
- Control Soup (Placebo Comparator): Negative control match for sodium (no MSG + 0.635% salt)
  Interventions: Dietary Supplement: Control soup no MSG

INTERVENTIONS:
Dietary Supplement: Soup with MSG — 0.5% MSG + 0.48% salt
  Arms: Soup with MSG
Dietary Supplement: Control soup no MSG — Negative control match for sodium (no MSG + 0.635% salt)
  Arms: Control Soup

SUMMARY:
The objective of this study is to compare energy intake following consumption 0.5% MSG versus a control with no added MSG and matched for sodium in healthy non-smoking premenopausal female adults.

DETAILED DESCRIPTION:
The study is a randomized, 2-arm, double-blind, placebo-controlled, Latin square cross-over clinical trial to assess the impact of 0.5% MSG on total and meal/snack-specific energy intake and on subjective ratings of appetite compared to sodium. Subjects will partake in an adaptation visit to avoid first order effects and will not be included in the randomization.

A total of 75 healthy premenopausal women aged 19 to 60 y (inclusive) will be randomized to a sequence of test product administration. Participants will consume 1 of 2 test products, based on randomization sequence at each test period visit. Carrot and coriander soup (0.5% MSG + 0.48% salt) or negative control match for sodium (no MSG + 0.635% salt).

Participants will be required to meet several inclusion and exclusion criteria, which will be assessed at the screening visit, including a health questionnaire, medical/medication history, eating behavior questionnaires, depression questionnaire and anthropometric measurements. After assessment of the eligibility criteria (see Eligibility section) at the screening visit, qualified participants will be invited to participate in the study and will be familiarized with the completion of VAS for subjective ratings of hunger, fullness, satiety and desire to eat.

Over a 3-week period, participants will come to the test facility on three occasions to complete the study with a one week wash-out period between each visit. Participants will fast overnight before each visit and consume the same evening meal before each test day.

Participants arrive at the research center at approximately 8:15am. Right before serving the breakfast meal, participants will be asked to complete a satiety rating questionnaire (using visual analogue scale (VAS)). At 8:30am, participants will consume breakfast (cereal and milk). Immediately after eating breakfast participants will complete another VAS questionnaire as well as a taste/liking meal evaluation. Thereafter, VAS will be completed at 30 minute intervals.

Four hours after the breakfast meal (at 12:30pm), participants will be given one of the test products (carrot and coriander soup with or without MSG) based on their randomization schedule. Subjects will have 10 min to consume the soup in its entirety. Following test product/soup intake, subjects will complete a taste/liking meal evaluation and VAS questionnaire. Immediately after completion of the questionnaire (12:40pm), an ad lib lunch buffet will be provided and participants will be instructed to eat as much as or as little as they desire (within 30 min) until comfortably full, followed by completing a taste/liking meal evaluation and VAS questionnaire. Thereafter, VAS will be completed at 30 minute intervals.

At 3:30pm, participants will be provided with their second portion of the test product to consume within 10 min, followed by completing a taste/liking meal evaluation and VAS questionnaire. Immediately after test soup administration and completing questionnaires, an ad lib snack buffet will be provided and participants will be instructed to eat as much as or as little as they desire within 20 min, followed by completing a taste/liking meal evaluation and VAS questionnaire. VAS assessment will continue at 30 min intervals thereafter until 5:00pm ending the study day. Participants' next visit will be scheduled after 1 week wash-out period: all procedures are identical with the exception of the test treatment soup consumed by participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Premenopausal Female, 19 to 60 yrs old
* Non-smoker
* Non-heavy Drinker
* BMI between 25 and 39.9 inclusive at the screening visit (with average BMI 30)
* no reported current or previous metabolic diseases or chronic gastrointestinal disorders
* no medically prescribed diet, no slimming diet, used to eating 3 meals a day and snacking
* No blood donation during the study
* Reported intense sporting activities ≤ 10h/w
* Reported alcohol consumption ≤14 units/w
* Informed consent signed
* Recruitment form filled out

Exclusion Criteria:

* Smoker
* Vegetarian
* Disliking the meals provided on the test day, have allergy or intolerance to test products or study meals
* Use of medication which interferes with study measurements (as judged by the study physician).
* Possible eating disorder (measured by SCOFF questionnaire score >1)
* Current depression measured by BDI <10
* Pregnant during the study period or in the six months prior to pre-study investigation
* Reported lactating 6 weeks before pre-study investigation and during the study
* Reported weight loss or gain ≥ 10 % of bodyweight during a period of six months before pre-study examination.
* Eating disorder (measured by SCOFF questionnaire, ≥2 "yes" responses)
* Reported participation in another biomedical trial 1 month before the start of the study

Ages: 19 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The difference in total energy intake (lunch and snack) compared with a control, as determined by food amount that subject consumed using a food scale (weigh foods before and after). | 8 hours 30 min Postprandial Study
  food will be measured before and after using a food scale (weight out and in)

SECONDARY OUTCOMES:
The difference in energy intake only at lunch compared with a control, as determined by food amount that subject consumed using a food scale (weigh foods before and after). | 8 hours 30 min Postprandial Study
  food will be measured before and after using a food scale (weight out and in)
The difference in energy intake of snack only compared with a control | 8 hours 30 min Postprandial Study
  food will be measured before and after using a food scale

OTHER OUTCOMES:
The difference in subjective feelings of appetite using visual analogue scales (VAS), compared with a negative control | 8 hours 30 min Postprandial Study
Taste meal evaluation, including soup liking | 8 hours 30 min Postprandial Study

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Pombo, PhD, Principal Investigator — Nutrition & Health Enquires, Leatherhead Food Research
Locations (1):
- Leatherhead Food Research, Leatherhead, Surrey, United Kingdom